CLINICAL TRIAL: NCT02495948
Title: One Month Clinical Comparison of Lotrafilcon B and Samfilcon A
Brief Title: Comparison of Two Marketed Silicone Hydrogel Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: CLA560-P001
Record Dates: First submitted 2015-07-09; First posted 2015-07-13 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors | interventions — Abortion, Induced

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AOA then ULTRA (Other): Lotrafilcon B contact lenses worn first, followed by samfilcon A contact lenses. Each product worn bilaterally (in both eyes) for a minimum of 5 days/week, 8 hours/day for 30 days in a daily wear modality.
  Interventions: Device: Lotrafilcon B contact lenses; Device: Samfilcon A contact lenses; Device: Hydrogen peroxide solution; Device: Saline solution
- ULTRA then AOA (Other): Samfilcon A contact lenses worn first, followed by lotrafilcon B contact lenses. Each product worn bilaterally for a minimum of 5 days/week, 8 hours/day for 30 days in a daily wear modality.
  Interventions: Device: Lotrafilcon B contact lenses; Device: Samfilcon A contact lenses; Device: Hydrogen peroxide solution; Device: Saline solution

INTERVENTIONS:
Device: Lotrafilcon B contact lenses
  Other Names: AIR OPTIX® AQUA
Device: Samfilcon A contact lenses
  Other Names: Bausch + Lomb ULTRA
Device: Hydrogen peroxide solution — Used as a cleaning, disinfection, and storage solution for silicone hydrogel and soft contact lenses
  Other Names: CLEAR CARE®
Device: Saline solution — Used for rinsing contact lenses, as needed
  Other Names: SENSITIVE EYES® PLUS

SUMMARY:
The purpose of this study is to evaluate cholesterol sorption by AIR OPTIX® AQUA lenses compared to ULTRA lenses after 30 days of wear.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent document;
* Vision correctable to 20/40 Snellen (feet) or better in each eye at distance with both study contact lenses;
* Willing to wear study lenses on a daily basis (minimum 5 days/week, 8 hours/day) and attend all study visits;
* Successful wear of single-vision spherical, 2-week/ monthly replacement silicone hydrogel contact lenses in both eyes daily wear during the past 2 months for a minimum of 5 days/week, 8 hours/day. (Note: Monovision is included);
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any anterior segment infection, inflammation, disease or abnormality that contraindicates contact lens wear (within 7 days of enrollment, or current);
* History of herpetic keratitis, corneal surgery or irregular cornea;
* Any use of systemic or ocular medications within the past 30 days for which contact lens wear could be contraindicated as determined by the investigator;
* Monocular (only 1 eye with functional vision) or fit with only one lens;
* Current or past AIR OPTIX® AQUA or ULTRA lens wearers;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Manager, Vision Care, GCRA, Study Director — Alcon, A Novartis Division

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 10 investigational sites located in the US.
Pre-assignment Details: Of the 168 enrolled, 1 participant was exited as a screen failure prior to randomization. This reporting group includes all randomized participants (167).
Period: Period 1, First 30 Days of Wear
Arm/Group | AOA Then ULTRA | ULTRA Then AOA
Started | 83 | 84
Completed | 83 | 83
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 2, Second 30 Days of Wear
Arm/Group | AOA Then ULTRA | ULTRA Then AOA
Started | 83 | 83
Completed | 82 | 82
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized participants (Intent-to-Treat (ITT) analysis set).
Groups:
- Overall: Lotrafilcon B and samfilcon A contact lenses worn during Period 1 and Period 2 in a crossover assignment, as randomized.
Arm/Group | Overall
Number analyzed (Participants) | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (9.01)
Gender [Count of Participants; unit: Participants]
  Female | 130
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Mean Ex-vivo Cholesterol Deposits After 30 Days of Wear
Description: The contact lens (right eye) was removed and stored dry and frozen until analysis. Total cholesterol deposits (cholesterol and cholesterol esters) were extracted from the lens and measured in micrograms. Lower deposits indicate increased lens performance. Study originally intended to analyze 36 lenses per arm, but actual number of lenses analyzed was less due to measurement error.
Time Frame: Day 30, each product
Population: Intent-to-Treat analysis set
Measure: Mean (Standard Deviation); unit: micrograms
Units Other Than Participants: Lenses
Groups:
- AIR OPTIX AQUA (AOA): Lotrafilcon B contact lenses worn during Period 1 or Period 2 for 30 days
- ULTRA: Samfilcon A contact lenses worn during Period 1 or Period 2 for 30 days
Arm/Group | AIR OPTIX AQUA (AOA) | ULTRA
Number analyzed (Participants) | 167 | 167
Number analyzed (Lenses) | 34 | 33
micrograms | 1.63 (2.21) | 4.89 (3.12)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of informed consent throughout the duration of a subject's participation in the study (at least 62 days). AEs are reported as pre-treatment and treatment-emergent. Ocular AEs are presented for both study eye and non-study eye combined.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the medical device.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to the initiation of study treatment
- AIR OPTIX AQUA: All subjects exposed to lotrafilcon B contact lenses during Period 1 or Period 2
- ULTRA: All subjects exposed to samfilcon A contact lenses during Period 1 or Period 2
Arm/Group | Pretreatment | AIR OPTIX AQUA | ULTRA
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/166 | 0/167
Other Adverse Events (participants affected / at risk) | 0/168 | 0/166 | 0/167

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.